CLINICAL TRIAL: NCT00470340
Title: Arterial LIPIODOLISED Chemotherapy Versus Systemic Chemotherapy With Gemcitabine Plus Oxaliplatin (GEMOX) Versus no Treatment Following Surgical Resection or Local Ablation of Hepatocellular Carcinoma in Cirrhotic Patients
Brief Title: Chemotherapy or Not, Following Complete Treatment of Hepatic Cancer in Cirrhotic Patients
Acronym: GEMOXIAL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: during the study
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Isabelle Brindel, Department of Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P051062
Record Dates: First submitted 2007-05-04; First posted 2007-05-07 (Estimated); Last update posted 2011-05-05 (Estimated); Status verified 2007-05

CONDITIONS: Liver Neoplasms; Liver Cirrhosis; Carcinoma, Hepatocellular; Recurrence; Neoplasm Recurrence, Local
Keywords: Recurrence; Neoplasm Recurrence, Local; Liver; Liver Neoplasms; Liver Cirrhosis; Carcinoma, Hepatocellular; Iodized Oil; gemcitabine [Substance Name]; oxaliplatin [Substance Name]; gemcitabine-oxaliplatin regimen [Substance Name]; Randomized Controlled Trials; Multicenter Studies; Cisplatin; Injections, Intra-Arterial; Injections, Intravenous; Chemotherapy, Adjuvant
MeSH Terms: conditions — Liver Neoplasms; Liver Cirrhosis; Carcinoma, Hepatocellular; Recurrence; Neoplasm Recurrence, Local | interventions — Oxaliplatin; Gemcitabine; Cisplatin; Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Oxaliplatin, gemcitabine, cisplatin, lipiodol
  Interventions: Drug: Oxaliplatin, gemcitabine, cisplatin, lipiodol
- 2 (Experimental): Oxaliplatin, gemcitabine, cisplatin, lipiodol
  Interventions: Drug: Oxaliplatin, gemcitabine, cisplatin, lipiodol

INTERVENTIONS:
Drug: Oxaliplatin, gemcitabine, cisplatin, lipiodol — Oxaliplatin, gemcitabine, cisplatin, lipiodol

SUMMARY:
Besides liver transplantation, the curative treatment of primary hepatic cancer with cirrhosis remains the surgical resection. Radiofrequency or cryotherapy currently allow local ablation of small cancer, with very good results. However, all these treatments are followed by high rates of recurrence (50 - 70% at 5 years). Then, it seems essential to associate to the surgical resection or to the local ablation as "adjuvant" treatment, in order to prevent or to decrease the rate of recurrence. However, no evidence supports this attitude. Therefore, following curative treatment of primary hepatic cancer with cirrhosis, we propose to compare treated to untreated patients. Postoperative treatment means either intra-arterial chemotherapy or systemic chemotherapy. The main criterion of the study is time of survival without recurrence. The main secondary objective is the safety.

DETAILED DESCRIPTION:
The best treatment for hepatocellular carcinoma (HCC) with cirrhosis, currently is liver transplantation because treating the cancer and the causal disease. For the majority of patients, transplantation is not proposed, and the curative treatment remains the surgical resection. Radiofrequency or cryotherapy currently allows local destruction (or ablation) of the small HCC, with results that seem equivalent to the surgical resection. These last techniques increase the therapeutic possibilities in the presence of hepatic insufficiency. However, all these treatments are followed by high rates of recurrence (50 - 70% at 5 years and close to 100% at 10 years). The development of tumoral nodules, undetected at the time of the curative treatment, or the occurrence of new HCC, under the effects of the cirrhotic process or viral genomic modifications explain these disappointing results. Therefore, it seems essential to associate an adjuvant treatment to the surgical resection or the local destruction. Intra-arterial chemotherapy with or without embolisation is a largely evaluated therapeutic approach whose results are contradictory. Several retrospective studies, seem nevertheless to show a benefit of this treatment in adjuvant situation. Systemic chemotherapy for a long time regarded as ineffective, currently has a renewed interest due to the use of new drugs like gemcitabine and oxaliplatin (GEMOX regimen). This regimen showed a certain effect in a phase II study in advanced forms of HCC with cirrhosis. We propose to test by a prospective randomized multicentric phase III study, the effectiveness of an adjuvant treatment by systemic chemotherapy or intra-arterial LIPIODOLISED chemotherapy (CIAL), after surgery or complete local destruction of HCC. Three groups will be compared: a group of untreated patients (n=109), a group of patients treated by intra-arterial chemotherapy (CIAL = cisplatin 75 mg + lipiodol 10 ml; 3 courses every 6 weeks)(n=77) and a group of patients treated by systemic chemotherapy (GEMOX= day 1: gemcitabine 1000 mg/m² iv within 100 min; day 2: oxaliplatin 100 mg/m² iv within 2h; 8 courses every 2 weeks, d1 = d14)(n=77). Selection and randomisation are planned 4-8 weeks following complete treatment of the HCC. Identical follow up for the 3 groups includes clinical, biological, morphological exams every 3 months for 2 years, then every 6 months for 3 years. The main criterion of the study is survival without recurrence. The secondary objectives are the global survival, the safety and an estimate of the costs of the various treatments. The awaited results are 1) to demonstrate the effectiveness of at least one of these adjuvant treatment following complete treatment of HCC in cirrhotic patients and 2) to determine the best adjuvant treatment. Estimated inclusion time is 2 years, with an analysis of the principal criterion at 3 years. Follow-up of 5 years is envisaged for each patient, leading to a 7 years duration study.

ELIGIBILITY:
Inclusion Criteria:

* Hepatocellular carcinoma (histology or Barcelona criteria) curatively treated by surgical resection or by radiofrequency or by cryotherapy
* Evidence of liver cirrhosis (clinical, biological, endoscopic or histological criteria)
* Morphological evaluation 4 to 6 weeks following curative treatment
* No evidence of local or distant disease on the morphological evaluation
* Absence of peritoneal or lymph node metastasis
* Absence of pre- or per-operative macroscopic tumoral thrombus
* Minimal free margin of 5 mm following pathological exam
* ALPHAAFOETOPROTEINE level of less than 4 normal values or decreased by 50%, 4 to 6 weeks following curative treatment
* Biological criteria, 2 weeks before treatment as follow:

  * neutrophilic polymorphonuclear > 1500/mm3,
  * platelets > 100 000/mm3,
  * total bilirubin < 25 mmol/l (1.46 mg/dl),
  * creatinin < 1.5 x normal value
* Eastern Cooperative Oncology Group (ECOG) equal to 0 or 1
* Life expectancy > 12 weeks
* Absence of sensitive neuropathy at inclusion time
* Health insurance coverage
* Efficient contraceptive method if applicable
* Signed informed consent

Exclusion Criteria:

* Curative treatment performed 10 weeks or more before the beginning of adjuvant treatment
* Contraindication to an angiography or hepatic artery thrombosis or portal thrombosis.
* Pregnant or breastfeeding woman
* Concomitant involvement to any clinical trial
* Decompensate cirrhosis and Child-Pugh score ≥ 8 or clinical ascitis.
* Cancer of the Liver Italian Program (C.L.I.P.) score ≥ 2
* Heart or lung insufficiency
* Other cancer not considered as definitively cured
* Creatinin clearance < 30 ml/min
* Recurrence of HCC less than 12 months following any last treatment
* Any radiotherapy during the 4 weeks before inclusion
* Known sensitivity to any drug of this protocol
* Immunodeficiency (HIV+, transplanted patient)
* Inability of follow up
* Impossibility of clear understanding of the protocol for no french speaking patient
* Patient under legal protection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 263 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Survival without recurrence at 2 years | 2 years

SECONDARY OUTCOMES:
Morbidity and mortality following adjuvant treatment | at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric Savier, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Urc La Pitie Salpetriere,, Poissy, France